CLINICAL TRIAL: NCT00333983
Title: Evaluation of Robotic Arm Rehabilitation in Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3833-R
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2014-03-20 (Estimated); Last update posted 2014-03-20 (Estimated); Status verified 2014-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Robot Exercise Group
  Interventions: Device: Robotic Upper Extremity Neurorehabilitation
- Arm 2 (Active Comparator): Traditional Upper Extremity Exercise Group
  Interventions: Other: Traditional Upper Extremity Exercise Group

INTERVENTIONS:
Device: Robotic Upper Extremity Neurorehabilitation — Upper extremity exercise using a planar robot Upper extremity exercise using a planar and vertical robot
  Arms: Arm 1
Other: Traditional Upper Extremity Exercise Group — Upper extremity stretching, skateboard reaching activities, and arm ergometer
  Arms: Arm 2

SUMMARY:
The purpose of this study is to compare 2 training programs using robotic exercise devices to supervised arm exercises in stroke patients with chronic stable deficits.

DETAILED DESCRIPTION:
A robotic exercise device has been developed(MIT-MANUS)capable of providing therapy to the arm for patients with weakness due to stroke. The randomized trial will compare conventional care, planar robot intervention and an intervention of planar and vertical robot training among patients with chronic, stable deficits. We will evaluate motor outcomes, effectiveness, cost, patient satisfaction and quality of life. The study will determine the efficacy of upper extremity robot therapy compared to supervised self-administered exercise therapy in patients with deficits due to stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a clinically, defined, unilateral, hemiparetic stroke with radiologic exclusion of other diagnoses
* Stroke onset greater than six months before randomization for ischemic stroke patients and one year before randomization for hemorrhagic stroke patients
* A grade 3 or lower in Manual Muscle Test in the hemiparetic elbow flexion and shoulder abduction

Exclusion Criteria:

* Subjects unable to give informed consent
* Serious complicating medical illness
* Contracture or orthopedic problems limiting the range of joint movement in the study arm
* Visual loss
* Stroke occurred within 6 months for ischemic stroke patients, one year for hemorrhagic patients
* Botox treatment within 3 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-06; Primary Completion 2010-04 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Bever, MD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Result] Conroy SS, Whitall J, Dipietro L, Jones-Lush LM, Zhan M, Finley MA, Wittenberg GF, Krebs HI, Bever CT. Effect of gravity on robot-assisted motor training after chronic stroke: a randomized trial. Arch Phys Med Rehabil. 2011 Nov;92(11):1754-61. doi: 10.1016/j.apmr.2011.06.016. Epub 2011 Aug 17. PMID 21849168

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 147 community-dwelling adults with a diagnosis of chronic stroke were referred for study criteria screening by local VA stroke clinics and PT/OT clinicians. Community study advertisements and flyers were also utulized during this recruitment period that started October 2006 and ended December 2009.
Pre-assignment Details: Participants were excluded prior to randomization if they did not meet inclusion/exclusion criteria. Some candidates declined after learning of the study length and schedule committment.
Groups:
- Planar Robot: Robot-assisted planar reaching x 60 minutes
- Planar + Vertical Robot: Robot-assisted planar and robot-assisted vertical reaching x 60 minutes
- Intensive Conventional Exercise: Upper extremity stretching, skateboard reaching activites, range of motion and arm ergometer x 60 minutes.
Period: Overall Study
Arm/Group | Planar Robot | Planar + Vertical Robot | Intensive Conventional Exercise
Started | 20 | 21 | 21
Completed | 17 | 16 | 19
Not Completed | 3 | 5 | 2
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intensive Conventional Exercise: Upper extremity stretching, skateboard reaching activities, range of motion, and arm ergometer training x 60 minutes.
- Total: Total of all reporting groups
Arm/Group | Planar Robot | Planar + Vertical Robot | Intensive Conventional Exercise | Total
Number analyzed (Participants) | 20 | 21 | 21 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 17 | 19 | 52
  >=65 years | 4 | 4 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (12) | 60 (13) | 56 (6.3) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 11 | 28
  Male | 12 | 12 | 10 | 34
Region of Enrollment [Number; unit: participants]
  United States | 20 | 21 | 21 | 62
Fugl-Meyer Upper Extremity Motor Assessment [Mean (Standard Deviation); unit: units on a scale] — The upper extremity portion of the Fugl-Meyer Motor Assessment has a range of 0 to 66 with 0 being the minimum score and 66 the maximum. A higher score indicates a better outcome.
  units on a scale | 20.3 (14.7) | 16.5 (10.6) | 18.2 (12.5) | 18.0 (12.5)

OUTCOME MEASURES:

1. Primary Outcome: Upper Extremity Portion of the Fugl-Meyer Motor Performance Assessment
Description: The Fugl-Meyer Assessment (FMA) is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia (Fugl-Meyer, Jaasko, Leyman, Olsson, & Steglind, 1975; Gladstone, Danells, & Black, 2002).
  Sections can be administered separately and the upper extremity motor portion of this measure was used as our primary outcome. Assessment items included movement, coordination, and reflex action of the shoulder, elbow, forearm, wrist, and hand. These items were scored on the basis of ability to complete using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully.
  The total possible score for the upper extremity is 66 with a minimum range of 0 and maximum of 66. A higher score indicates a better outcome.
Time Frame: Baseline to Final Training (6 weeks)
Population: The number of participants analyzed were based on an intention to treat methodology with the exception of individuals that were non-compliant with the protocol or did not progress to the midpoint (3 week) evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Planar Robot: Planar Robot Exercise x 60 minutes.
- Planar + Vertical: Planar + Vertical Robot Exercise x 60 minutes.
Arm/Group | Planar Robot | Planar + Vertical | Intensive Conventional Exercise
Number analyzed (Participants) | 20 | 21 | 21
units on a scale | 3.27 (3.27) | 2.51 (3.33) | 1.82 (4.24)
Statistical Analysis 1: Comparison: Planar Robot vs Planar + Vertical vs Intensive Conventional Exercise; An analysis of all robot interventions compared with intensive conventional exercise for Fugl-Meyer change were completed using linear mixed models; Test type: Superiority or Other; p = .025, Mixed Models Analysis — P value was set at .025 to adjust for 2 treatment comparisons and for interim monitoring for the treatment effect

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 6 month time period for each participant which included baseline testing, intervention and retention.
Groups:
- Planar Robot: Planar Robot Exercise Group
- Planar + Vertical Robot: Planar + Vertical Robot Exercise Group
- Intensive Conventional Exercise: Upper extremity stretching, skateboard reaching activities, range of motion and arm ergometer training.
Arm/Group | Planar Robot | Planar + Vertical Robot | Intensive Conventional Exercise
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 2/20 | 1/21 | 1/21
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Planar Robot (N=20) | Planar + Vertical Robot (N=21) | Intensive Conventional Exercise (N=21)
Hospitalization (General disorders) | 2 (2) | 1 (1) | 0 (0) — One participant experienced non-study related renal failure. One participant experienced non-study related medical status change. One participant experienced non-study related hip fracture after fall at home.
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) — One participant with shouler pain in the study arm limiting participation in traditional upper extremity exercise.

LIMITATIONS AND CAVEATS:
This study was terminated early with the current number of subjects analyzed. A midstudy futility analysis showed a need for 99 participants per group to determine signifcance between the robotic training over the intensive conventional exercise.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes